CLINICAL TRIAL: NCT05466019
Title: Toripalimab Combined With FLOT Regimen for Perioperative Treatment of PD-L1 Positive Locally Advanced Resectable Gastric Cancer or Gastroesophageal Junction Adenocarcinoma (GEJ): a Prospective, Single-center Clinical Study
Brief Title: A Prospective, Single Center Clinical Study of Toripalimab Combined With FLOT Regimen for Perioperative Treatment of PD-L1 Positive Locally Advanced Resectable Gastric Cancer or Gastroesophageal Junction Adenocarcinoma (GEJ)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, Professor, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARS-GC04
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: PD-L1 Positive Locally Advanced Patients With Resectable Gastric Cancer
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toripalimab combined with FLOT regimen (Experimental): The enrolled patients will receive 3 cycles of FLOT regimen +Toripalimab treatment before surgery, and every 2 weeks is a treatment cycle (Q2W). After completing the 3 cycles of treatment, the patient undergoes surgical resection.Toripalimab combined with FLOT regimen were maintained for 4 cycles after surgery.
  Interventions: Drug: Drug: Toripalimab, FLOT(Docetaxel+oxaliplatin+leucovorin+5-FU)

INTERVENTIONS:
Drug: Drug: Toripalimab, FLOT(Docetaxel+oxaliplatin+leucovorin+5-FU) — FLOT: Docetaxel 50mg/m2 ivd d1 + oxaliplatin 85mg/m2 ivd d1 + leucovorin 200mg/m2 ivd d1 + 5-FU 2600mg/m2 civ, Q2W Toripalimab 3mg/kg, intravenously administered on the first day of each cycle, Q2W.

SUMMARY:
In this study, patients with PD-L1 positive locally advanced patients with resectable gastric cancer or gastroesophageal junction adenocarcinoma were invited to participate in the study.To evaluate the efficacy and safety of patients with PD-L1 positive gastric cancer or gastroesophageal junction adenocarcinoma (≥T3 and the number of lymph node metastasis ≥1, and No distant metastasis) using Toripalimab combined with docetaxel, oxaliplatin, fluorouracil, leucovorin (FLOT regimen) .

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of the patient;
2. 18 years old <age <75 years old;
3. The researcher judged that he could comply with the study protocol;
4. Histologically confirmed gastric or gastroesophageal junction adenocarcinoma (Siewert II-III);
5. Clinical stage at admission: ≥T3 with ≥1 lymph node metastasis and no distant metastasis (AJCC 8th)

   * Esophagogastroduodenoscopy must be performed
   * Diagnostic laparoscopy must be performed
6. Immunohistochemistry confirmed that the patient was PD-L1 positive (CPS≥1);
7. Preoperative ECOG [Using the ECOG scoring standard Zubrod-ECOG-WHO (ZPS, 5-point method) developed by the Eastern Cooperative Oncology Group (ECOG)] Physical State Score 0/1;
8. Preoperative ASA score I-III;
9. Expected survival ≥12 weeks;
10. The baseline blood routine and biochemical parameters of selected patients should meet the following criteria:

    * Hemoglobin ≥90g/ L, which can be met by blood transfusion;
    * Absolute neutrophil count ≥1.5×10^9/ L
    * Platelet count ≥100×10^9/ L
    * Aspartic acid or alanine aminotransferase ≤ 2.5 times the upper limit
    * Alkaline phosphatase ≤ 2.5 times normal upper limit (ULN),
    * Thyroid stimulating hormone (TSH) ≤1 times ULN (if abnormal, T3 and T4 levels should be investigated at the same time; if T3 and T4 levels are normal, they can be included in the group);

Exclusion Criteria:

1. Inestigators identified stage IV (metastatic) or unresectable gastric or gastroesophageal junction adenocarcinoma
2. Previous systemic treatment for gastric cancer
3. Have a history of allergy to any component of terriprizumab, oxaliplatin, capecitabine;
4. Received any of the following medical treatment:

   A. Have received anti-PD-1 or anti-PD-L1 antibody therapy in the past; B. Have received any investigational drug treatment within 4 weeks before using the drug for the first time; C. Enroll in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up; D. Receive the last dose of anti-cancer treatment (including radiotherapy) within 4 weeks before the first use of the study drug;; E. Receive systematic treatment with corticosteroids (> 10mg prednisone equivalent daily dose) or other immunosuppressants within 2 weeks prior to their first use of the study drug; F. Those who have been vaccinated with anti-tumor vaccines or the study drugs have been vaccinated with live vaccines within 4 weeks before the first administration; G. Those who have undergone major surgery or trauma within 4 weeks before using the study drug for the first time;
5. History of other malignant diseases within 5 years;
6. History of active autoimmune disease or autoimmune disease
7. The subject has cardiovascular clinical symptoms or disease that is not well controlled;
8. Severe infection 4 weeks prior to first use of study drug (CTCAE > Level 2)
9. A history of interstitial lung disease (except for radiation pneumonia not treated with Chinese hormone) or non-infectious pneumonia;
10. Patients with active pulmonary tuberculosis infection found by history or CT examination, or patients with active pulmonary tuberculosis infection history within 1 year before enrollment, or patients with active pulmonary tuberculosis interference history more than 1 year ago but without formal treatment;
11. Pregnant or lactating women;
12. Suffering from severe mental illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | 3 months

SECONDARY OUTCOMES:
event-free survival (EFS) | 2 years
disease-free survival (DFS) | 2 years
overall survival (OS) | 2 years
objective response rate (ORR) | 3 months
R0 Surgical conversion rate | 3 months
major pathological response (MPR) | 3 months
Incidence and severity of adverse events | 6 months
index of tumor-infiltrating lymphocyte (sTIL) infiltration | 3 months
type and number of intestinal flora | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China